CLINICAL TRIAL: NCT05609409
Title: FlexED: A Digital, Gamified Early Intervention for Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Cyprus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00111571
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Eating Disorders; Body Image
Keywords: Eating Disorders; Body Image Flexibility; Acceptance and Commitment Therapy; Psychological Flexibility; Online; Early Intervention
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Noncurrent Multiple Baseline Experimental Design where subjects will serve as their own control.
  Participants will be randomized to different baseline durations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Intervention (Experimental): Eight 20-30 minute sessions of an online, multimedia application
  Interventions: Behavioral: FlexED

INTERVENTIONS:
Behavioral: FlexED — Intervention consists of eight 20-30 minute sessions of a digital intervention based on Acceptance and Commitment Therapy (ACT). Participants learn skills of body image flexibility by following an avatar through a story line and completing interactive exercises.

SUMMARY:
The goal of this multiple baseline experiment is to test the effect of a digital, gamified early intervention for eating disorders on body image flexibility and determine treatment dose. Twenty-four young women and girls (between the ages of 15-25) with eating disorder (ED) symptoms will be randomized to different baseline durations (varying between 2-6 weeks). Participants will complete eight 20-30 minute sessions of a multimedia application over 10 weeks using their home computer or mobile device. Body Image Flexibility (BIF) will be measured repeatedly using a multimodal assessment strategy (behavior, physiological and self-report) during baseline and treatment phases. The investigators will estimate the effect of the intervention on BIF and examine when change occurs and plateaus (with no discernable benefit for additional sessions) to determine treatment dose.

ELIGIBILITY:
Inclusion Criteria:

* Female identified 15-25 years old
* Weight Concerns Scale score of >47
* Maladaptive weight control behaviors with onset <3 years

Exclusion Criteria:

* Currently meets full diagnostic criteria anorexia or bulimia nervosa or has in the past.
* Psychosis, substance use disorder or current suicidal ideation or self-harm.
* Start or change in psychiatric medications within the past month.
* NonEnglish Speaking.
* Presents with other specified feeding or eating disorder (OSFED) that does not have weight/shape concerns as a primary feature (e.g., Avoidant Restrictive Food Intake Disorder).

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female-identified
Enrollment: 34 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Change in body image flexibility as indexed by the Body Image - Acceptance and Action Questionnaire-5 (BI-AAQ-5) | Baseline, 1, 2, 3, 4, 6, 8, 10, 12, and 16 weeks
  5-item measure assessing the ability to behave flexibly in the presence of negative thoughts and feelings about the body. Scores range from 5 to 35 with higher scores indicating greater flexibility.
Change in High Frequency Heart Rate Variability (HF-HRV) | Baseline, 1, 2, 3, 4, 6, 8, 10, 12, and 16 weeks
  Heart rate variability during provocation of body image distress; greater variability indicates an increased capacity to modulate arousal and distress.
Change in biased processing of body image stimuli relative to neutral stimuli | Baseline, 1, 2, 3, 4, 6, 8, 10, 12, and 16 weeks
  Biased processing of stimuli is assessed using an emotional Stroop task with body image and neutral stimuli. Improvements are indicated by changes in reaction time and fewer errors.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT05609409/ICF_000.pdf